CLINICAL TRIAL: NCT05899010
Title: A Phase III Randomized Controlled Trial Comparing the Efficacy, Safety and Tolerability of Two Formulations of Vaginal Micronized Progesterone
Brief Title: MIcronized PROgesterone in Frozen Embryo Transfer Cycles
Acronym: MI-PROF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-MIC-2022-03; 2022-001045-21 (EudraCT Number)
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal progesterone 600mg (Active Comparator): Vaginal progesterone 600mg daily (200mg tid) will be started and maintained until 10 weeks of pregnancy or either up to menses or up to negative pregnancy test performed 10 days after ET
  Interventions: Drug: Vaginal progesterone 600mg daily
- Vaginal progesterone 800mg (Experimental): Vaginal progesterone 800mg daily (400mg bid) will be started and maintained until 10 weeks of pregnancy or either up to menses or up to negative pregnancy test performed 10 days after ET.
  Interventions: Drug: Vaginal progesterone 800mg daily

INTERVENTIONS:
Drug: Vaginal progesterone 600mg daily — If endometrial thickness (ETH) ≥7 mm and follicle dominance/ultrasound (US) signs of ovulation P levels are measured: if P ≤1.5 patients start LPS, else cycle is cancelled. If ETH <7mm and no follicle dominance: estradiol dose is increased to 9mg/day and new US is performed up to 4 days after. If persistent thin endometrium after dose increase, cycle is cancelled. 24-48h pre ET, E2 and P are measured. in the morning, pre VMP dose, or at least 6h after last progesterone dose. If progesterone <10ng/ml, additional 300mg daily oral micronized progesterone is administered on the day of the ET and maintained until 10 weeks pregnancy or up to menses or up to negative pregnancy test 10 days after ET. ET will be performed with available blastocysts 6 days after start of LPS. 3-5 days, after ET, a blood test for P measurement will be performed in the morning, before VMP dose, or at least 6h after last progesterone dose. 10 days after ET, the last P test will be done with pregnancy test.
  Arms: Vaginal progesterone 600mg
Drug: Vaginal progesterone 800mg daily — If endometrial thickness (ETH) ≥7 mm and follicle dominance/ultrasound (US) signs of ovulation P levels are measured: if P ≤1.5 patients start LPS, else cycle is cancelled. If ETH <7mm and no follicle dominance: estradiol dose is increased to 9mg/day and new US is performed up to 4 days after. If persistent thin endometrium after dose increase, cycle is cancelled. 24-48h pre ET, E2 and P are measured. in the morning, pre VMP dose, or at least 6h after last progesterone dose. If progesterone <10ng/ml, additional 300mg daily oral micronized progesterone is administered on the day of the ET and maintained until 10 weeks pregnancy or up to menses or up to negative pregnancy test 10 days after ET. ET will be performed with available blastocysts 6 days after start of LPS. 3-5 days, after ET, a blood test for P measurement will be performed in the morning, before VMP dose, or at least 6h after last progesterone dose. 10 days after ET, the last P test will be done with pregnancy test.
  Arms: Vaginal progesterone 800mg

SUMMARY:
This randomized trial was designed as non-inferiority trial aiming to compare ongoing pregnancy rates following LPS with 600 mg/day vs 800 mg/day vaginal VMP. All patients will undergo an artificial cycle frozen embryo transfer (AC-FET) with transdermal estradiol 6mg/day Patients undergoing an artificial cycle FET will start estrogen priming with transdermal estradiol 6mg/day (Estrogel®) on cycle D1-D3. Following 10-12 days of estrogen priming, patients will be randomized to luteal phase support with a standard formulation (200mg tid, Utrogestan®) or a new formulation (400mg bid) VMP. All patients will undergo a serum P measurement on the day before embryo transfer (ET). Patients with P<10 ng/ml will receive a supplement of oral micronized progesterone 300mg, while patients with P≥10ng/ml will maintain the previous luteal phase support (LPS) protocol

ELIGIBILITY:
Inclusion Criteria:

* Endometrial preparation with hormone replacement therapy
* Age 18-43 years following an autologous IVF cycle (with or without preimplantation genetic testing for aneuploidy)
* Age < 50 years following an egg donation cycle
* BMI > 18 and < 30 kg/m2
* blastocyst embryo transfer
* Willing to participate in the study
* Able to come to the Center to comply with the procedures of the study: blood tests, appointments and drug dispensation.

Exlusion Criteria:

* • Uterine diseases (e.g. submucosal fibroids, polyps, previously diagnosed Müllerian abnormalities)
* Hydrosalpinx
* Recurrent pregnancy loss (≥ 3 previous miscarriages)
* Recurrent implantation failure (≥ 3 previously failed embryo transfers of good-quality blastocysts)
* Allergy to study medication
* Pregnancy or lactation
* Contraindication for hormonal treatment
* Personalized initiation of exogenous progesterone according to a previous endometrial receptivity assay test
* Recent history of severe disease requiring regular treatment (clinically significant concurrent medical condition that could compromise subject safety or interfere with the trial assessment).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1020 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 7-9 weeks after embryo transfer
  A positive heart beat at ultrasound after 11-13 weeks of gestation

SECONDARY OUTCOMES:
Implantation rate | 3-4 weeks after embryo transfer
  Number of gestational sacs over total embryo transfered
Biochemical pregnancy rate | 10 to 12 days after embryo transfer
  positive beta-human chorionic gonadotropin (hCG)
Clinical pregnancy rate | 3-4 weeks after embryo transfer
  A positive heart beat at ultrasound
Miscarriage rate | before completion of 12 weeks of gestation
  any spontaneous abortion that occurred after confirmation of clinical pregnancy
Frequency of adverse events | Until 15 days after the end of treatment with progesterone

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD, PhD, Study Chair — Service of Reproductive Medicine Dexeus University Hospital; Noemie Sachs-Guedj, MD, Principal Investigator — Service of Reproductive Medicine Dexeus University Hospital
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Geyter C, Calhaz-Jorge C, Kupka MS, Wyns C, Mocanu E, Motrenko T, Scaravelli G, Smeenk J, Vidakovic S, Goossens V; European IVF-monitoring Consortium (EIM) for the European Society of Human Reproduction and Embryology (ESHRE). ART in Europe, 2015: results generated from European registries by ESHRE. Hum Reprod Open. 2020 Feb 24;2020(1):hoz038. doi: 10.1093/hropen/hoz038. eCollection 2020. PMID 32123753
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Background] Shi Y, Sun Y, Hao C, Zhang H, Wei D, Zhang Y, Zhu Y, Deng X, Qi X, Li H, Ma X, Ren H, Wang Y, Zhang D, Wang B, Liu F, Wu Q, Wang Z, Bai H, Li Y, Zhou Y, Sun M, Liu H, Li J, Zhang L, Chen X, Zhang S, Sun X, Legro RS, Chen ZJ. Transfer of Fresh versus Frozen Embryos in Ovulatory Women. N Engl J Med. 2018 Jan 11;378(2):126-136. doi: 10.1056/NEJMoa1705334. PMID 29320646
- [Background] Wei D, Liu JY, Sun Y, Shi Y, Zhang B, Liu JQ, Tan J, Liang X, Cao Y, Wang Z, Qin Y, Zhao H, Zhou Y, Ren H, Hao G, Ling X, Zhao J, Zhang Y, Qi X, Zhang L, Deng X, Chen X, Zhu Y, Wang X, Tian LF, Lv Q, Ma X, Zhang H, Legro RS, Chen ZJ. Frozen versus fresh single blastocyst transfer in ovulatory women: a multicentre, randomised controlled trial. Lancet. 2019 Mar 30;393(10178):1310-1318. doi: 10.1016/S0140-6736(18)32843-5. Epub 2019 Feb 28. PMID 30827784
- [Background] Roque M, Haahr T, Geber S, Esteves SC, Humaidan P. Fresh versus elective frozen embryo transfer in IVF/ICSI cycles: a systematic review and meta-analysis of reproductive outcomes. Hum Reprod Update. 2019 Jan 1;25(1):2-14. doi: 10.1093/humupd/dmy033. PMID 30388233
- [Background] Groenewoud ER, Cohlen BJ, Al-Oraiby A, Brinkhuis EA, Broekmans FJ, de Bruin JP, van den Dool G, Fleisher K, Friederich J, Goddijn M, Hoek A, Hoozemans DA, Kaaijk EM, Koks CA, Laven JS, van der Linden PJ, Manger AP, Slappendel E, Spinder T, Kollen BJ, Macklon NS. A randomized controlled, non-inferiority trial of modified natural versus artificial cycle for cryo-thawed embryo transfer. Hum Reprod. 2016 Jul;31(7):1483-92. doi: 10.1093/humrep/dew120. Epub 2016 May 13. PMID 27179265
- [Background] Ghobara T, Gelbaya TA, Ayeleke RO. Cycle regimens for frozen-thawed embryo transfer. Cochrane Database Syst Rev. 2017 Jul 5;7(7):CD003414. doi: 10.1002/14651858.CD003414.pub3. PMID 28675921
- [Background] Groenewoud ER, Cohlen BJ, Macklon NS. Programming the endometrium for deferred transfer of cryopreserved embryos: hormone replacement versus modified natural cycles. Fertil Steril. 2018 May;109(5):768-774. doi: 10.1016/j.fertnstert.2018.02.135. PMID 29778369
- [Background] Vaisbuch E, de Ziegler D, Leong M, Weissman A, Shoham Z. Luteal-phase support in assisted reproduction treatment: real-life practices reported worldwide by an updated website-based survey. Reprod Biomed Online. 2014 Mar;28(3):330-5. doi: 10.1016/j.rbmo.2013.10.022. Epub 2013 Nov 14. PMID 24447959
- [Background] Nawroth F, Ludwig M. What is the 'ideal' duration of progesterone supplementation before the transfer of cryopreserved-thawed embryos in estrogen/progesterone replacement protocols? Hum Reprod. 2005 May;20(5):1127-34. doi: 10.1093/humrep/deh762. Epub 2005 Feb 3. PMID 15695314
- [Background] Griesinger G, Blockeel C, Sukhikh GT, Patki A, Dhorepatil B, Yang DZ, Chen ZJ, Kahler E, Pexman-Fieth C, Tournaye H. Oral dydrogesterone versus intravaginal micronized progesterone gel for luteal phase support in IVF: a randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2212-2221. doi: 10.1093/humrep/dey306. PMID 30304457
- See also: Related Info — http://www.dexeus.com